CLINICAL TRIAL: NCT01265160
Title: Jiangzhuo Prescription ，Fenofibrate and Placebo in the Treatment of Hyperlipidemia (Syndrome of Phlegm Obstruction)Clinical Study (JZF)
Acronym: JZF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Other Study IDs: 81929
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Last update posted 2010-12-23 (Estimated); Status verified 2010-09

CONDITIONS: Metabolic Syndromes; Hyperlipidemia
MeSH Terms: conditions — Metabolic Syndrome; Hyperlipidemias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- the group of Jiangzhuo prescription
- the group of fenofibrate
- the group of placebo

SUMMARY:
Jiangzhuo prescription ,fenofibrate and placebo in the treatment of hyperlipidemia(syndrome of phlegm obstruction), randomized, parallel-controlled, multi-center clinical study

DETAILED DESCRIPTION:
Charged by the five research centers in line with traditional Chinese medicine syndrome of phlegm obstruction 240 cases have hyperlipidemia, and overweight, as well as hypertension or diabetes were randomly divided into Chinese herbal compound Jiangzhuo prescription group and western medicine fenofibrate group and placebo group.The treatment groups were compared 12-week regulation of blood lipids and step-down, blood sugar effect.

ELIGIBILITY:
Inclusion Criteria:

* 1. Consistent with diagnosed hyperlipidemia, TG≥2.26mmol/L and ≤7.0mmol/L. 2. Aged 18-65 years old. 3.BMI ≥ 24kg/m2, but <35 kg/m2. 4. Waist circumference ≥ 90cm (male) or waist circumference ≥ 80cm (women). 5. Comply with any of the following 3 :bloode pressure elevated levels of:SBP ≥130mmHg or DBP ≥85mmHg; fasting plasma glucose (FPG) increased: FPG ≥ 100mg/dl (5.6mmol / l ), or previously diagnosed type 2 diabetes or have received appropriate treatment.

Exclusion Criteria:

* 1. Has been used to control lipidsdrugs, but use the time for those below the 3 month.

  2.Secondary dyslipidemia, such as nephrotic syndrome, hyperthyroidism, etc. 3.Taking thyroid medications and other drugs that affect lipid metabolism, such as high-dose thiazide diuretics, β-receptor blockers, corticosteroids.

  4.Severe diseases of heart, lung, liver, kidney, brain, blood ,etc. 5.With the treatment of insulin, sulfonylureas, rosiglitazone or metformin. 6.3 months prior to the study of myocardial infarction or unstable angina confirmed.

  7.Uncontrolled blood sugar or after controlling FPG>7.0mmol/L or 2hPG>11.1mmol/L 8.Uncontrolled blood pressure or after contraolling blood pressure>140/90mmHg 9.ALT≥80mmol/L 10.Pregnancy, for pregnancy or breast-feeding women 11.Allergis of fibrates or Chinese medicine 12.Mental illness 13.Cancer patients 14.History of gallbladder disease or cholelithiasis 15.With the treatment of Cyclosporine or coumarin anticoagulants 16.The patient with other clinical studies in the past 3 months 17.History of alcoholism and drug dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Combined metabolic syndrome in patients with hyperlipidemia
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-05 (Estimated); Study Completion 2011-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beijing Chinese Medicine Hospital, Beijing
  - Beijing Ji Shui Tan Hospital, Beijing
  - Beijing Medical University,DONGZHIMEN Hospital, Beijing
  - Civil Aviation General Hospital, Beijing